CLINICAL TRIAL: NCT05941039
Title: Effects of Vestibular Training on Postural Control of Healthy Adults Using Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clarkson University (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Kwadwo Appiah-Kubi, Assistant Professor of Physical Therapy, Clarkson University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-25
Record Dates: First submitted 2023-03-23; First posted 2023-07-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality; Vestibular Training; Balance Assessment
Keywords: VR; Balance; Vestibular Training; EMG; EOG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vestibular Activation Training (Experimental)
  Interventions: Device: Vestibular training using VR followed by Control; Device: Control followed by Vestibular training using VR
- No Training (No Intervention)

INTERVENTIONS:
Device: Vestibular training using VR followed by Control — A cross-over design will be used with group one receiving the training intervention for 6 days, a 4-day washout period, and a 6-day no-training period.
  Arms: Vestibular Activation Training
Device: Control followed by Vestibular training using VR — Group two will follow the reverse sequence.
  Arms: Vestibular Activation Training

SUMMARY:
Postural instability is a common symptom of vestibular dysfunction that impacts a person's day-to-day activities. Vestibular rehabilitation is effective in decreasing dizziness, visual symptoms and improving postural control through several mechanisms including sensory reweighting. As part of the sensory reweighting mechanisms, vestibular activation training with headshake activities influence vestibular reflexes. However, combining challenging vestibular and postural tasks to facilitate more effective rehabilitation outcomes is under-utilized. The novel concurrent headshake and weight shift training (Concurrent HS-WST) is purported to train the vestibular system to directly impact the postural control system simultaneously and engage sensory reweighting to improve balance. Young healthy participants will perform the training by donning a virtual reality headset with an overhead harness on and a spotter present to prevent any falls. The investigators propose that this training strategy would show improved outcomes over traditional training methods by improving vestibular-ocular reflex (VOR) gains, eye movement variability, sensory reweighting and promoting postural balance. The findings of this study may guide clinicians to develop rehabilitation methods for vestibular postural control in neurological populations with vestibular and/or sensorimotor control impairment.

ELIGIBILITY:
Inclusion Criteria:

* Able to stand independently (without an assistive device)
* This study requires participants to perform postural assessments including reactive balance following mechanical perturbations.
* Participants will also perform headshake activities and weight shift training in standing for 20 mins will mini breaks.
* Participants must be within the age of 18-35.
* A power analysis revealed that a sample of 24 participants will required for a two-group comparison to detect a significant difference at alpha=0.05 and 0.30 effect size at beta=0.8 (G*Power, Version 3.0.10)(Faul et al, 2007).

Exclusion Criteria:

* Participants with an evidence of:
* Concussion, vestibular, balance or oculomotor issues for the prior 6 months.
* Neuropathic conditions, particularly affecting the lower extremities. Participants with this issue will have sensory impairments which can affect their sensory assessment.
* Current musculoskeletal deficits including significant postural abnormalities (signs of spinal, pelvic and leg length discrepancies).
* Pain or limitations in neck range of motion.
* Recent (within 6 months) orthopedic surgery that impacts postural training.
* Visual Impairment
* Participants must be able to see and follow targets on the computer monitor. Therefore, subjects must have 20/50 (corrected) vision. Subjects who are blind cannot participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Vestibulo-ocular reflex (VOR) gain | Two week study period
  Horizontal and vertical vestibulo-ocular reflex (VOR) gain will be assessed using the video head impulse test (vHIT; ICS, Otometrics, Taastrup, Denmark). Twenty head impulses each will be performed to assess each direction of the semicircular canals with participant in a seated position
Eye movement variability | Two week study period
  Horizontal and vertical eye movements will be assessed during force plate perturbation trials using BlueGain electro-oculography (EOG) device (Cambridge Research Systems). Participants will stand on a force plate perturbation device with EOG electrodes affixed on eye muscles to record eye movements during toes up (simulating being pushed backward) and toes down (simulating being pushed forward) perturbation rotation trials.
Electromyography (EMG) amplitude | Two week study period
  Electromyography (EMG) will be assessed during force plate perturbation trials using Delsys Trigno wireless sensors (Delsys Inc., Boston, MA). Participants will stand on a force plate perturbation device with EMG sensors placed on postural muscles to record electrical activity during toes up (simulating being pushed backward) and toes down (simulating being pushed forward) perturbation rotation trials.
Electromyography (EMG) time onset | Two week study period
  Electromyography (EMG) will be assessed during force plate perturbation trials using Delsys Trigno wireless sensors (Delsys Inc., Boston, MA). Participants will stand on a force plate perturbation device with EMG sensors placed on postural muscles to record electrical activity during toes up (simulating being pushed backward) and toes down (simulating being pushed forward) perturbation rotation trials.
Balance equilibrium and composite scores | Two week study period
  Equilibrium and composite scores will be assessed by the Modified Clinical Test for Sensory Interaction on Balance (MCTSIB; NeuroCom®, Natus Medical Inc., Pleasanton, CA) during quiet stance. The MCTSIB requires the participant to stand upright as stable as possible for 10 s under four different conditions: (1) eyes open (EO) on a stable surface (SS), (2) eyes closed (EC) on SS, (3) EO on foam surface (FS), (4) EC on FS.
Sensory ratios | Two week study period
  Sensory ratios will be assessed by the Modified Clinical Test for Sensory Interaction on Balance (MCTSIB; NeuroCom®, Natus Medical Inc., Pleasanton, CA) during quiet stance. The MCTSIB requires the participant to stand upright as stable as possible for 10 s under four different conditions: (1) eyes open (EO) on a stable surface (SS), (2) eyes closed (EC) on SS, (3) EO on foam surface (FS), (4) EC on FS.

CONTACTS AND LOCATIONS:
Locations (1):
- Clarkson University, Potsdam, New York, United States

REFERENCES:
- [Background] Appiah-Kubi KO, Wright WG. Vestibular training promotes adaptation of multisensory integration in postural control. Gait Posture. 2019 Sep;73:215-220. doi: 10.1016/j.gaitpost.2019.07.197. Epub 2019 Jul 16. PMID 31376748